CLINICAL TRIAL: NCT07164196
Title: Evaluation of Angiopoietin-like Protein 4 Levels in Patients With Endometriosis
Brief Title: Endometriosis-Angiopoietin-like Protein-4
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Merve Didem Eşkin Tanrıverdi, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: TABED 1-25-1372
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Angiopoietin-like Protein-4; Pelvic Pain
Keywords: Endometriosis; Angiopoietin-like protein-4; Peritoneal fluid; Inflammation
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Inflammation | interventions — Angiopoietin-Like Protein 4; CA-125 Antigen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples were collected through antecubital venous blood sampling. In the study group, serum samples were obtained just before laparoscopy, while peritoneal fluid (PF) samples were collected from the Douglas pouch during trocar insertion into the abdominal cavity. Serum and PF levels of Angiopoietin-like protein-4 were analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis group (Study group): The study group included women with endometriosis. The study group consisted of women diagnosed with endometriosis who consecutively underwent laparoscopic endometriosis surgery.
  Interventions: Other: Angiopoietin-like protein-4 (ANGPTL4) Peritoneal Fluid Level; Other: Cancer Antigen 125 (CA-125) Serum Level; Other: Angiopoietin-like protein-4 (ANGPTL4) Serum Level
- Healthy women (Control group): Control group consisted of healthy women. The control group consisted of women who consecutively visited the outpatient clinic for routine gynecologic examinations and had no known diseases.
  Interventions: Other: Cancer Antigen 125 (CA-125) Serum Level; Other: Angiopoietin-like protein-4 (ANGPTL4) Serum Level

INTERVENTIONS:
Other: Angiopoietin-like protein-4 (ANGPTL4) Peritoneal Fluid Level — Measurement of peritoneal fluid levels of Angiopoietin-like protein-4 (ANGPTL4) level by ELISA method.
  Groups: Endometriosis group (Study group)
Other: Cancer Antigen 125 (CA-125) Serum Level — Measurement of venous blood serum level of CA-125 level by ELISA method.
Other: Angiopoietin-like protein-4 (ANGPTL4) Serum Level — Measurement of venous blood serum level of Angiopoietin-like protein-4 (ANGPTL4) Level level by ELISA method.

SUMMARY:
Endometriosis is a chronic inflammatory disease associated with pelvic pain, dyspareunia, and impaired ovarian reserve. Cancer antigen-125 (CA-125) is widely studied but limited by low specificity, while angiopoietin-like protein-4 (ANGPTL4) has emerged as a potential biomarker due to its role in angiogenesis and inflammation. In the current study it was aimed to investigate serum and peritoneal fluid ANGPTL4 levels in women with endometriosis compared to healthy controls, and to evaluate their associations with clinical symptoms, serum CA-125, and anti-Müllerian hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometriosis for study group who underwent laparoscopic endometriosis surgery
* Healthy women for control group

Exclusion Criteria:

* Cardiovascular diseases including hypertension
* Type 1 or type 2 diabetes mellitus
* Morbid obesity
* Primary adrenal insufficiency
* Uterine fibroids
* Thyroid dysfunctions including Hashimoto thyroiditis and Grave's disease
* Hepatic dysfunctions
* Renal insufficiency
* Genetic disorders in chromosome constitution or karyotype analysis including monosomy X, trisomy X and gene mutations as BMP15, FMR I, POFIB, and GDF9
* Neurologic diseases
* Psychiatric disorders
* Autoimmune diseases or syndromes including Addison's disease, autoimmune syndromes, scleroderma, Sjogren's syndrome, myasthenia gravis, inflammatory bowel diseases, multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus and familial Mediterranean fever
* History of any malignancy
* History of exposure to chemotherapeutic agents or radiotherapy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Endometriosis is characterized by the presence of endometrial tissue outside the uterus, including the ovaries, fallopian tubes, peritoneal membrane, or abdominal cavity, and it is diagnosed exclusively in females.
Study Population: Study population includes a total of 80 participants. The study group consists of 40 women with the diagnosis of endometriosis, and the control group consists of 40 healthy women.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Serum and peritoneal fluid Angiopoietin-like protein-4 level | day 1
  Nanogram/milliliter

SECONDARY OUTCOMES:
Serum cancer antigen 125 level | day 1
  Unit/milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Merve Didem Eşkin Tanrıverdi, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Not Valid, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD are available which may be shared in necessary conditions.

REFERENCES:
- [Background] Campara K, Rodrigues P, Viero FT, da Silva B, Trevisan G. A systematic review and meta-analysis of advanced oxidative protein products levels (AOPP) levels in endometriosis: Association with disease stage and clinical implications. Eur J Pharmacol. 2025 Jun 5;996:177434. doi: 10.1016/j.ejphar.2025.177434. Epub 2025 Feb 28. PMID 40024324
- [Background] Makoui MH, Fekri S, Makoui RH, Ansari N, Esmaeilzadeh A. The Role of Mast Cells in the Development and Advancement of Endometriosis. Am J Reprod Immunol. 2025 Mar;93(3):e70019. doi: 10.1111/aji.70019. PMID 40028674
- [Background] Falcone T, Flyckt R. Clinical Management of Endometriosis. Obstet Gynecol. 2018 Mar;131(3):557-571. doi: 10.1097/AOG.0000000000002469. PMID 29420391
- [Background] Brown R, Imran SA, Wilkinson M. Lipopolysaccharide (LPS) stimulates adipokine and socs3 gene expression in mouse brain and pituitary gland in vivo, and in N-1 hypothalamic neurons in vitro. J Neuroimmunol. 2009 Apr 30;209(1-2):96-103. doi: 10.1016/j.jneuroim.2009.02.001. Epub 2009 Mar 3. PMID 19261336